CLINICAL TRIAL: NCT05262647
Title: A Prospective Study for Effectiveness of 18F-FAPI PET in the Diagnosis of Liver Fibrosis: Comparison With Liver Biopsy
Brief Title: 18F-FAPI PET in the Diagnosis of Liver Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Other Study IDs: QYFYWZLL26714
Record Dates: First submitted 2021-12-15; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Liver Fibrosis; FAP; Positron Emission Tomography
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: 18F-FAPI — Patients with chronic liver disease underwent 18F-FAPI-04 PET/CT and percutaneous liver biopsy.

SUMMARY:
It is an open label observation clinical trial, all participants are chronic liver disease. The investigators deem to make a novel evaluate criteria to hepatic fibrosis. The point of the clinical trial is to evaluate the novel biomaker 18F-FAPI-04 by PET-CT scan in the evaluation of the hepatic fibrosis.

DETAILED DESCRIPTION:
Participants are with clinically confirmed chronic liver disease,including chronic viral hepatitis, autoimmune hepatitis, liver disease after liver transplantation, nonalcoholic fatty liver disease, alcoholic hepatitis, primary biliary cholangitis, primary sclerosing cholangitis and congestive hepatopathy etc.

Participants are without liver tumor and other liver disease besides liver fibrosis Participants has no history of malignant tumors Participants agree to performe FAPI PET and liver biopsy

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed chronic liver disease,including chronic viral hepatitis, autoimmune hepatitis, liver disease after liver transplantation, nonalcoholic fatty liver disease, alcoholic hepatitis, primary biliary cholangitis, primary sclerosing cholangitis and congestive hepatopathy etc.
* Without liver tumor and other liver disease besides liver fibrosis
* No history of malignant tumors
* Agree to performe FAPI PET and liver biopsy

Exclusion Criteria:

* Pregnancy
* With anti-hepatic fibrosis treatment in 6 months
* With contraindications to percutaneous liver biopsy,for such as uncooperative patient, severe coagulopathy, extrahepatic biliary obstruction,etc.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients has been pathological diagnosis as Liver Fibrosis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-12-12 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
18F-FAPI PET in the Diagnosis of Liver Fibrosis | 12.01.2021 to12.01.2022
  18F-FAPI as a PET-CT biomarker to Liver Fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Guangjie Yang, PhD, Study Chair — The affiliated hostpital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, Shandong, China